CLINICAL TRIAL: NCT01599598
Title: Coherence Training for Military Personnel
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: United States Naval Medical Center, San Diego (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NMCSD.2011.0130
Record Dates: First submitted 2012-05-07; First posted 2012-05-16 (Estimated); Last update posted 2016-08-19 (Estimated); Status verified 2016-08

CONDITIONS: Stress
Keywords: perceived stress; depression; anxiety; posttraumatic stress disorder; military; school; training environment; heart rate variability; progressive muscle relaxation; psychophysiological coherence; coherence advantage; stress reduction; stress regulation; independent duty corpsmen
MeSH Terms: conditions — Depression; Anxiety Disorders; Stress Disorders, Post-Traumatic | interventions — Autogenic Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Progressive Muscle Relaxation (Active Comparator): A stress intervention where subjects will learn to regulate stress based on the tensing and releasing of the major muscle groups in the body, accompanied with relaxed breathing techniques.
  Interventions: Behavioral: Progressive Muscle Relaxation
- Coherence Advantage (Active Comparator): A stress intervention where subjects will learn to regulate stress by focusing on breathing and mindfulness techniques while recognizing physiological coherence by way of a portable biofeedback device.
  Interventions: Behavioral: Coherence Advantage

INTERVENTIONS:
Behavioral: Progressive Muscle Relaxation — Participants will be instructed to practice the techniques twice daily for 5-15 minutes per session, and subsequently use the techniques when confronted with a stressful event such as a project deadline, exam, skill evaluation, etc. Participants in this condition will listen to PMR instruction by way of a mp3 player.
  Arms: Progressive Muscle Relaxation
Behavioral: Coherence Advantage — Participants will be instructed to practice the techniques twice daily for 5-15 minutes per session, and subsequently use the techniques when confronted with a stressful event such as a project deadline, exam, skill evaluation, etc. Participants in this condition will practice the techniques while using a biofeedback device to recognize when they enter psychophysiological coherence.
  Other Names: emWave2
  Arms: Coherence Advantage

SUMMARY:
Military operations and training situations present many physical and psychological challenges for service members to adapt to and overcome. The challenges of these changing conditions necessitate having to cope with stress, which is seen as the negative perceptions, feelings, and emotions that manifest from the subjective physical and/or mental strain on life processes. In addition, service members are returning from deployments having gone through traumatic experiences that can develop into posttraumatic stress disorder (PTSD), depression or other serious conditions. The Surface Warfare Independent Duty Corpsman (IDC) School is an example of a training environment where some students may be entering the program with symptoms of PTSD, which may preclude or make it more difficult for them to perform well. Autonomic nervous system (ANS) dysregulation has been observed in patients with PTSD and those experiencing chronic stress, such that there is more arousing, sympathetic input to the heart than calming, parasympathetic input, which is usually the dominant division of the ANS involved in controlling one's heart rate. The IDC training program is an example of an environment where the service member is expected to excel while being subjected to multiple sources of stress. The fast tempo coupled with performance expectations may induce stress and actually inhibit learning. The Institute of HeartMath has developed the Coherence Advantage program which teaches one to self-regulate their emotions while focusing on breathing to compliment the active process of self-regulation. In conjunction, the emWave Personal Stress Reliever allows the user to receive heart rate variability (HRV) biofeedback, hence giving the user the opportunity to self-regulate their ANS through breathing and self-regulation techniques. The proposed study will test the effectiveness of the Coherence Advantage program versus progressive muscle relaxation (PMR) in reducing stress symptomatology among Surface Warfare IDC students. The effectiveness of these two different interventions will be compared on outcomes of PTSD, depression, anxiety, sleep quality, perceived stress, attrition, and class performance.

ELIGIBILITY:
Inclusion Criteria:

* Sailors
* Enrolled as students in the Surface Warfare Medicine Institute's Independent Duty Corpsman School

Exclusion Criteria:

* Administratively rolled over into another class
* Dropped out of the school (due to academic or medical reasons)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2012-04; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Stress symptomatology | 12 months
  The effectiveness of the two stress intervention trainings will be evaluated on symptoms of depression, posttraumatic stress disorder, generalized anxiety, perceived stress, and sleep quality.

SECONDARY OUTCOMES:
School performance | 12 months
  The effectiveness of the two stress intervention trainings will be evaluated on final grades.
Attrition | 12 months
  The effectiveness of the two stress intervention trainings will be evaluated on rates of attrition.

CONTACTS AND LOCATIONS:
Overall Officials: Scott L Johnston, PhD, Principal Investigator — U.S. Navy, Medical Service Corps, Naval Center for Combat & Operational Stress Control (NCCOSC)
Locations (1):
- Surface Warfare Medicine Institute, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No